CLINICAL TRIAL: NCT04153292
Title: SAPIEN M3 System Transcatheter Mitral Valve Replacement Via Transseptal Access
Brief Title: The ENCIRCLE Trial
Acronym: ENCIRCLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-19
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Mitral Regurgitation; Mitral Valve Insufficiency
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- TMVR - Main Cohort (Experimental): Subjects for whom commercially available surgical or transcatheter treatment options are deemed unsuitable will have transcatheter mitral valve replacement (TMVR).
  Interventions: Device: SAPIEN M3 valve and dock
- TMVR - Failed TEER Registry (Experimental): Subjects who have had an attempted but failed transcatheter edge-to-edge repair (TEER) procedure will have TMVR.
  Interventions: Device: SAPIEN M3 valve and dock
- TMVR - MAC Registry (Experimental): Subjects with mitral annular calcification (MAC) will have TMVR.
  Interventions: Device: SAPIEN M3 valve and dock

INTERVENTIONS:
Device: SAPIEN M3 valve and dock — During the procedure a SAPIEN M3 dock and a SAPIEN M3 valve will be implanted via transseptal approach.

SUMMARY:
This study will establish the safety and effectiveness of the SAPIEN M3 System in subjects with symptomatic, at least 3+ mitral regurgitation (MR) for whom commercially available surgical or transcatheter treatment options are deemed unsuitable.

Following completion of enrollment, subjects will be eligible for enrollment in the continued access phase of the trial.

DETAILED DESCRIPTION:
This is a prospective single-arm, multicenter study.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. MR ≥ 3+
3. NYHA functional class ≥ II
4. Per the Heart Team, commercially available surgical or transcatheter treatment options are deemed unsuitable due to clinical, anatomic or technical considerations.
5. Subject's heart failure management has been optimized based on subject characteristics and applicable guidelines, and stable for at least 30 days prior to enrollment.
6. The subject or subject's legal representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent.

Exclusion Criteria:

1. Mitral/cardiac anatomy that would preclude appropriate delivery and deployment of the SAPIEN M3 dock or valve
2. Inappropriate anatomy for femoral introduction and delivery of the SAPIEN M3 dock and valve
3. Presence of any device that will contact or interfere with the SAPIEN M3 System during delivery or after implantation
4. Left ventricular ejection fraction <25%
5. Severe right ventricular dysfunction
6. Need for aortic, tricuspid or pulmonic valve intervention within the next 12 months
7. History of heart transplant
8. Cardiac imaging evidence of intracardiac mass, thrombus or vegetation
9. Active bacterial endocarditis within 180 days of the procedure
10. Hemodynamic instability requiring inotropic or mechanical support within 30 days of the procedure
11. Myocardial infarction within 30 days of the procedure
12. Clinically significant untreated coronary artery disease requiring revascularization
13. Any percutaneous cardiovascular intervention, cardiovascular surgery, or carotid surgery within 30 days of the procedure
14. Stroke or transient ischemic attack within 90 days of the procedure
15. Irreversible, severe pulmonary hypertension
16. Chronic obstructive pulmonary disease requiring home oxygen therapy or chronic outpatient oral steroid use
17. Renal insufficiency or receiving renal replacement therapy
18. Liver disease
19. Planned surgery within the next 12 months
20. Inability to tolerate or a medical condition precluding treatment with antithrombotic therapy, including heparin administration during the procedure
21. Active infection requiring current antibiotic therapy
22. Active SARS-CoV-2 infection (Coronavirus-19 [COVID-19]) or previously diagnosed with COVID-19 with sequelae that could confound endpoint assessments
23. Leukopenia, anemia, thrombocytopenia, history of bleeding diathesis or coagulopathy or hypercoagulable states
24. Refusal of blood products
25. Female who is pregnant or lactating
26. Estimated life expectancy <12 months due to non-cardiac conditions
27. Participating in another investigational drug or device study that has not reached its primary endpoint
28. Subject considered to be part of a vulnerable population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2031-02-28 (Estimated)

PRIMARY OUTCOMES:
Non-hierarchical composite of death and heart failure rehospitalization | 1 year
  Number of subjects with death and/or heart failure rehospitalization

SECONDARY OUTCOMES:
Improvement in NYHA functional class compared to baseline | 1 year
  New York Heart Association (NYHA) functional classification of heart failure is based on how much a patient is limited during physical activity. The rating ranges from I-IV. I = no limitations of physical activity; II = slight limitations of physical activity, ordinary physical activity results in fatigue, palpitation, shortness of breath; III = marked limitations of physical activity, less than ordinary activity causes fatigue, palpitation, or shortness of breath; IV = unable to carry on any physical activity without discomfort, symptoms of heart failure at rest.
Improvement in KCCQ Overall Score compared to baseline | 1 year
  The Kansas City Cardiomyopathy Questionnaire (KCCQ) is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. An overall summary score can be derived from the physical function, symptom (frequency and severity), social function and quality of life domains. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Improvement in MR compared to baseline | 1 year
  Number of subjects with improved MR compared to baseline
Decrease in LVEDVi compared to baseline | 1 year
  Number of subjects with decreased left ventricular end-diastolic volume index (LVEDVi) compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: John Webb, MD, Principal Investigator — St. Paul's Hospital; Mayra Guerrero, MD, Principal Investigator — Mayo Clinic; David Daniels, MD, Principal Investigator — California Pacific Medical Center
Locations (68):
- United States (56):
  - Heart Center Hospital, Huntsville, Alabama
  - Banner University Medical Center, Phoenix, Arizona
  - Saint Josephs Hospital Medical Center Dignity Health, Phoenix, Arizona
  - TMC Healthcare, Tucson, Arizona
  - Scripps Health, La Jolla, California
  - Good Samaritan Hospital, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Kaiser Sunset LA, Los Angeles, California
  - Saint Joseph Hospital, Orange, California
  - California Pacific Medical Center, San Francisco, California
  - UC Health Northern Colorado (Medical Center of the Rockies), Loveland, Colorado
  - Delray Medical Center, Delray Beach, Florida
  - Cardiac & Vascular Institute Foundation, Gainesville, Florida
  - Ascension St. Vincent's Hospital, Jacksonville, Florida
  - Naples Community Hospital, Naples, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Emory University, Atlanta, Georgia
  - Piedmont Healthcare, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Northshore University Health System, Glenview, Illinois
  - St. Vincent Heart Center of Indiana, Indianapolis, Indiana
  - University of Kansas, Kansas City, Kansas
  - Cardiovascular Research Institute of Kansas (CRIOK), Wichita, Kansas
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - Medstar Union Memorial Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's, Boston, Massachusetts
  - Henry Ford, Detroit, Michigan
  - Minneapolis Heart, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - CentraCare, Saint Cloud, Minnesota
  - Saint Luke's Kansas City, Kansas City, Missouri
  - St. Patrick Hospital, Missoula, Montana
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Morristown Medical Center, Morristown, New Jersey
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - University of Buffalo, Buffalo, New York
  - Weill Cornell Medicine, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Novant Health and Vascular Institute, Charlotte, North Carolina
  - The Christ Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - UPMC Heart and Vascular Institute, Mechanicsburg, Pennsylvania
  - Alleghany General Hospital, Pittsburgh, Pennsylvania
  - Saint Thomas Health, Nashville, Tennessee
  - Austin Heart, Austin, Texas
  - HCA Houston Healthcare Medical (SCRI), Houston, Texas
  - UT Memorial Hermann, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - Sentara Norfolk, Norfolk, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - University of Washington Seattle, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Australia (2):
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Prince Alfred Hospital, Camperdown
- Canada (3):
  - Laval University, Québec, Quebec
  - St. Michael's, Toronto
  - St. Pauls, Vancouver
- Israel (3):
  - Shaare Zedek Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Rotterdam Erasmus MC, Rotterdam
- United Kingdom (2):
  - Saint Bartholomew's Medical Center, London
  - Saint Thomas Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guerrero ME, Daniels DV, Makkar RR, Thourani VH, Asch FM, Pham M, Muhammad KI, Greenbaum AB, Vasquez A, Oldemeyer JB, Dahle TG, Rihal C, Morse MA, Rodriguez E, O'Neill BP, Russo M, Whisenant B, Yadav P, Yu X, Wang DD, Makar M, Baran DA, Mahoney P, Reddy G, Blanke P, Webb J; ENCIRCLE Trial Executive Committee and Study Investigators. Percutaneous transcatheter valve replacement in individuals with mitral regurgitation unsuitable for surgery or transcatheter edge-to-edge repair: a prospective, multicountry, single-arm trial. Lancet. 2025 Nov 29;406(10519):2541-2550. doi: 10.1016/S0140-6736(25)02073-2. Epub 2025 Oct 27. PMID 41167201